CLINICAL TRIAL: NCT00249769
Title: Assessment of the Non-Inferiority of the Concurrent Administration of Japanese Encephalitis Live Attenuated SA 14-14-2 Vaccine and Measles Vaccine Given Alone
Brief Title: Determining Safety and Efficacy of Japanese Encephalitis Vaccine When Given With Measles Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Research Institute for Tropical Medicine, Manila, Philippines (Unknown); Quintiles, Inc. (Industry); Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JEV01
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2018-09

CONDITIONS: Encephalitis, Japanese B
Keywords: Japanese Encephalitis; Japanese B Encephalitis; Japanese B Viral Encephalitis; Viral Encephalitis, Japanese B
MeSH Terms: conditions — Encephalitis, Japanese | interventions — Measles Vaccine

ARMS (3):
- LJEV then MV (Experimental): Received one dose of Live Japanese encephalitis vaccine SA 14-14-2 (LJEV) at 8 months of age, and one dose of measles vaccine (MV) one month later.
  Interventions: Biological: Live Japanese encephalitis vaccine SA 14-14-2 (LJEV); Biological: Measles Vaccine (MV)
- LJEV and MV (Experimental): Received one dose of Live Japanese encephalitis vaccine SA 14-14-2 (LJEV) concurrently with one dose of measles vaccine (MV) at 9 months of age.
  Interventions: Biological: Live Japanese encephalitis vaccine SA 14-14-2 (LJEV); Biological: Measles Vaccine (MV)
- MV then LJEV (Experimental): Received one dose of measles vaccine (MV) at 9 months of age, followed by one dose of Live Japanese encephalitis vaccine SA 14-14-2 (LJEV) one month later.
  Interventions: Biological: Live Japanese encephalitis vaccine SA 14-14-2 (LJEV); Biological: Measles Vaccine (MV)

INTERVENTIONS:
Biological: Live Japanese encephalitis vaccine SA 14-14-2 (LJEV) — Live Japanese encephalitis vaccine SA 14-14-2 (LJEV) is lyophilized powder that looks like a milky-white crisp cake. After reconstitution, it turns into a transparent orange red liquid. Its container is a vial. It is stored and transported between 2°C to 8°C and protected from light. Each single human dose is 0.5 ml containing not less than 5.4 log particle flux unit (PFU) of live Japanese Encephalitis (JE) virus. The 0.5ml injection is delivered subcutaneously via auto-disable syringe. Lot number 200411129-3 manufactured by Chengdu Institute of Biological Products (CDIBP), Chengdu, China.
Biological: Measles Vaccine (MV) — The Serum Institute of India (SII) measles vaccine provided routinely in the Expanded Program on Immunization (EPI) of the Philippines was the measles vaccine provided to the study participants. The vaccine met the requirements of the World Health Organization (WHO).
  SII measles vaccine contained live attenuated (freeze-dried) Edmonston-Zagreb strain measles virus propagated on human diploid cells (HDC). Each single human dose when reconstituted in a volume of 0.5 ml contains no less than 1000 Cell culture infectious dose 50% (CCID50) of live virus particles. SII measles vaccine is presented as a yellowish-white dry cake. The vaccine should be reconstituted with the diluent supplied (sterile water for injection). A sterile disposable syringe and needle are supplied separately. The 0.5ml injection is delivered subcutaneously via auto-disable syringe. Lot number 2979.

SUMMARY:
This study will determine whether it is safe and effective to administer Japanese encephalitis (JE) live attenuated SA 14-14-2 vaccine at the same time as measles vaccine. If it is found to be safe, it will pave the way for use in routine vaccination programs. The hypothesis is that children who receive JE live attenuated SA 14-14-2 vaccine and measles vaccine at the same time are protected against these diseases at the same level as those who receive the vaccines at different intervals.

DETAILED DESCRIPTION:
Japanese encephalitis is the leading cause of viral neurological disease and disability in Asia. The severity of sequelae, together with the volume of cases, make JE the most important cause of viral encephalitis in the world. Approximately 3 billion people-including 700 million children-live in Asian areas at risk for JE. JE most commonly infects children between the ages of 1 and 15 years, and can also infect adults in areas where the virus is newly introduced. More than 50,000 cases are reported annually and cause an estimated 10,000 to 15,000 deaths. This figure is believed to represent only a small proportion of the disease burden that actually exists.

An effective vaccine has existed since 1941, but has not reached the poorest countries in Asia. During the 60 years that the vaccine has been available, JE has infected an estimated 10.5 million children, resulting in more than 3 million deaths and more than 4 million children living with long-term disabilities. Control of this disease has been limited due to poor disease surveillance, a limited and unstable vaccine supply, lack of guidance and programmatic support for immunization, and limited advocacy.

A successful vaccine should be safe, efficacious, affordable, administered in a single dose, and easily incorporated into the routine Expanded Programmes on Immunization (EPI) programs. This study will help ensure the safety of SA 14-14-2 simultaneously administered with measles vaccine, paving the way for its use in routine EPI programs. If this candidate becomes widely available, it will drastically increase the feasibility of routine JE immunization in Asia, reducing the devastating death and disability caused by this disease. In addition to impacting low-income countries, the vaccine will allow countries that purchase vaccine-such as Thailand, Vietnam, Sri Lanka, and India-to recover health care dollars, improve their present programs, and address other unmet health care needs.

ELIGIBILITY:
Inclusion Criteria:

* Participant is healthy, aged between 8 months (± 2 weeks) at inclusion visit
* Subject is a full-term infant
* Subject's parents or legal guardian willing to provide signed informed consent.
* Children have completed 3 doses each of diphtheria, tetanus, pertussis (DTP) and oral polio vaccine (OPV).

Exclusion Criteria:

* History of documented HIV.
* Known or suspected impairment of immunologic function.
* History of serious chronic disease
* Underlying medical condition such as inborn errors of metabolism, failure to thrive, bronchopulmonary dysplasia, or any major congenital abnormalities requiring surgery or chronic treatment.
* Acute medical illness with or without fever within the last 72 hours or an axillary temperature ≥ 37.5°C at the time of inclusion.
* History of documented suspected encephalitis, encephalopathy, or meningitis
* History of measles
* History of thrombocytopenic purpura.
* Received any JE or measles vaccine prior to enrollment.
* Received any vaccine, other than the study vaccines, within 2 weeks prior to or scheduled to receive a non-study vaccination during the conduct of this trial.
* Hypotonic - hyporesponsiveness, after the preceding vaccination.
* History of seizures, including history of febrile seizures, or any other neurologic disorder.
* Prior or anticipated receipt of immune globulin or other blood products, or injected or oral corticosteroids or other immune modulator therapy except routine vaccines within 6 weeks of administration of the study vaccines. Individuals on a tapering dose schedule of oral steroids lasting <7 days may be included in the trial as long as they have not received more than one course within the last 2 weeks prior to enrollment.
* Suspected or known hypersensitivity to any of the investigational or marketed vaccine components.
* Serious adverse event related to the vaccine (i.e., possible, probably, definite)
* Persistent inconsolable crying (>3 hours) observed after a previous dose.
* Unable to attend the scheduled visits or comply with the study procedures.
* Enrolled in another clinical trial involving any therapy.
* Any condition that in the opinion of the investigator, would pose a health risk to the participant, or interfere with the evaluation of the study objectives.

Ages: 8 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2005-11-21 (Actual); Primary Completion 2006-05-30 (Actual); Study Completion 2006-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salvacion Gatchalian, MD, Principal Investigator — Research Institute for Tropical Medicine
Locations (1):
- Research Institute for Tropical Medicine, Manila, Philippines

REFERENCES:
- [Result] Gatchalian S, Yao Y, Zhou B, Zhang L, Yoksan S, Kelly K, Neuzil KM, Yaich M, Jacobson J. Comparison of the immunogenicity and safety of measles vaccine administered alone or with live, attenuated Japanese encephalitis SA 14-14-2 vaccine in Philippine infants. Vaccine. 2008 Apr 24;26(18):2234-41. doi: 10.1016/j.vaccine.2008.02.042. Epub 2008 Mar 18. PMID 18394765

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LJEV Then MV | LJEV and MV | MV Then LJEV
Started | 100 | 250 | 250
Received LJEV (Live Japanese encephalitis vaccine (LJEV)) | 100 | 236 | 224
Received Measles Vaccine | 97 | 236 | 235
Completed | 98 | 235 | 222
Not Completed | 2 | 15 | 28
Not completed — Withdrawal by Subject | 1 | 10 | 6
Not completed — Migration from Study Area | 1 | 3 | 14
Not completed — Miscellaneous | 0 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: The Safety population included all participants who received at least 1 vaccination.
Groups:
- Total: Total of all reporting groups
Arm/Group | LJEV Then MV | LJEV and MV | MV Then LJEV | Total
Number analyzed (Participants) | 100 | 236 | 235 | 571
Age, Continuous [Mean (Standard Deviation); unit: months] | 7.9 (0.3) | 8.9 (0.3) | 8.9 (0.3) | 8.7 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 108 | 128 | 284
  Male | 52 | 128 | 107 | 287
Weight [Mean (Standard Deviation); unit: kilograms] | 7.9 (1.0) | 8.0 (1.0) | 8.1 (1.0) | 8.0 (1.0)
Height [Mean (Standard Deviation); unit: centimeters] | 66.3 (2.6) | 67.6 (2.7) | 67.7 (2.6) | 67.4 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Seroprotection for Measles 4 Weeks After Vaccination
Description: Seroprotection after measles vaccination was defined as a measles antibody titer ≥ 120 mIU/mL. Measles immunoglobulin G (IgG) antibody was determined using the Enzygnost® Anti-Measles Virus/IgG enzyme-linked immunosorbent assay(ELISA) assay from Siemens, Marburg, Germany.
Time Frame: Day 0 (before vaccination) and Day 28 (4 weeks after measles vaccination)
Population: The per-protocol population includes randomized participants who received at least one vaccine dose excluding participants who did not meet the inclusion/exclusion criteria or were found non-compliant to the immunization or blood sampling schedule. The analysis includes participants with valid serology results for measles antibody during retesting.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LJEV Then MV | LJEV and MV | MV Then LJEV
Number analyzed (Participants) | 88 | 219 | 178
percentage of participants
  Day 0 | 1.1 [0.0 to 6.2] | 0.0 [0.0 to 1.7] | 0.0 [0.0 to 2.1]
  Day 28 | 88.6 [80.1 to 94.4] | 91.8 [87.3 to 95.1] | 86.5 [80.6 to 91.2]

2. Secondary Outcome: Percentage of Participants With Seroprotection for Japanese Encephalitis 4 Weeks After Vaccination
Description: Seroprotection after LJEV was defined as at least 1:10 dilution as recommended by the World Health Organization (WHO). JE antibody titers were determined by a plaque reduction neutralization test (PRNT).
Time Frame: Day 0 (before vaccination) and Day 28 (4 weeks after LJEV vaccination)
Population: Per protocol population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LJEV Then MV | LJEV and MV | MV Then LJEV
Number analyzed (Participants) | 88 | 222 | 180
percentage of participants
  Day 0 | 3.4 [0.7 to 9.6] | 5.4 [2.8 to 9.3] | 6.1 [3.1 to 10.7]
  Day 28 | 92.1 [84.3 to 96.7] | 90.5 [85.9 to 94.1] | 90.6 [85.3 to 94.4]

3. Secondary Outcome: Geometric Mean Concentration (GMC) of Measles Antibodies After Vaccination
Description: Measured using the Enzygnost® Anti-Measles Virus/IgG ELISA assay from Siemens, Marburg, Germany.
Time Frame: Day 0 (before vaccination) and Day 28 (4 weeks after measles vaccination)
Population: Per-protocol population; the analysis includes participants with valid serology results for measles antibody during retesting.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | LJEV Then MV | LJEV and MV | MV Then LJEV
Number analyzed (Participants) | 88 | 219 | 178
mIU/mL
  Day 0 | 12.8 [10.2 to 16.2] | 7.4 [6.3 to 8.8] | 7.0 [5.8 to 8.5]
  Day 28 | 318.9 [273.0 to 372.6] | 301.9 [269.0 to 338.9] | 262.5 [222.2 to 310.2]

4. Secondary Outcome: Geometric Mean Titer (GMT) of Japanese Encephalitis Antibodies After Vaccination
Description: Assayed by plaque reduction neutralization test (PRNT).
Time Frame: Day 0 (before vaccination) and Day 28 (4 weeks after LJEV vaccination)
Population: Per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | LJEV Then MV | LJEV and MV | MV Then LJEV
Number analyzed (Participants) | 88 | 219 | 178
titer
  Day 0 | 5.7 [4.9 to 6.5] | 5.7 [5.2 to 6.1] | 5.9 [5.3 to 6.6]
  Day 28 | 202.8 [140.5 to 292.9] | 155.0 [123.5 to 194.5] | 139.4 [109.5 to 177.5]

5. Secondary Outcome: Number of Participants Experiencing Local and Systemic Reactogenicity After Receiving Live Attenuated Japanese Encephalitis Vaccine (LJEV)
Description: Local reactions included erythema, pain, swelling, or induration. Systemic reactions included loss of appetite, crying, diarrhea, drowsiness, insomnia, irritability, vomiting, or fever. The parents of the participants recorded all local reactions and systemic events on an individual safety diary form.
Time Frame: Up to 7 days after LJEV administration
Population: Participants who received LJEV
Measure: Count of Participants; unit: Participants
Arm/Group | LJEV Then MV | LJEV and MV | MV Then LJEV
Number analyzed (Participants) | 100 | 236 | 224
Participants
  Local reactions: any | 27 | 53 | 27
  Local reactions: mild | 19 | 48 | 22
  Local reactions: moderate | 8 | 5 | 5
  Local reactions: severe | 0 | 0 | 0
  Systemic reactions: any | 58 | 97 | 88
  Systemic reaction: mild | 34 | 53 | 56
  Systemic reaction: moderate | 22 | 37 | 30
  Systemic reaction: severe | 2 | 7 | 2
  Fever: any | 24 | 52 | 57
  Fever: 37.5-38.6°C | 18 | 38 | 47
  Fever: 38.7-39.9°C | 6 | 14 | 10
  Fever: ≥ 40°C | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Experiencing Local and Systemic Reactogenicity After Receiving Measles Vaccine
Description: Local reactions included erythema, pain, swelling, and induration. Systemic reactions included loss of appetite, crying, diarrhea, drowsiness, insomnia, irritability, and vomiting. The parents of the participants recorded all local reactions and systemic events on an individual safety diary form.
Time Frame: Up to 7 days after measles vaccination
Population: Participants who received measles vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | LJEV Then MV | LJEV and MV | MV Then LJEV
Number analyzed (Participants) | 97 | 236 | 235
Participants
  Local reactions: any | 19 | 44 | 61
  Local reactions: mild | 15 | 42 | 50
  Local reactions: moderate | 4 | 2 | 11
  Local reactions: severe | 0 | 0 | 0
  Systemic reactions: any | 49 | 97 | 122
  Systemic reaction: mild | 31 | 53 | 77
  Systemic reaction: moderate | 13 | 37 | 42
  Systemic reaction: severe | 5 | 7 | 3
  Fever: any | 31 | 52 | 64
  Fever: 37.5-38.6°C | 21 | 38 | 52
  Fever: 38.7-39.9°C | 10 | 14 | 12
  Fever: ≥ 40°C | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Experiencing Unsolicited Adverse Events (AE)
Time Frame: Up to 7 days post-vaccination
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | LJEV Then MV | LJEV and MV | MV Then LJEV
Number analyzed (Participants) | 100 | 236 | 235
Participants
  Any Adverse Event | 35 | 43 | 79
  Related adverse event | 0 | 4 | 2
  Serious adverse event | 2 | 0 | 3

ADVERSE EVENTS:
Time Frame: 1 month for serious adverse events and 7 days for non-serious adverse events
Arm/Group | LJEV Then MV | LJEV and MV | MV Then LJEV
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/236 | 0/235
Serious Adverse Events (participants affected / at risk) | 5/100 | 0/236 | 7/235
Other Adverse Events (participants affected / at risk) | 34/100 | 43/236 | 78/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LJEV Then MV (N=100) | LJEV and MV (N=236) | MV Then LJEV (N=235)
Amoebiasis (Gastrointestinal disorders) | 1 | 0 | 2
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Urinary tract infection (Renal and urinary disorders) | 1 | 0 | 1
Acute Gastroenteritis (Gastrointestinal disorders) | 2 | 0 | 1
Bronchial Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Complex Febrile Seizure (Nervous system disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LJEV Then MV (N=100) | LJEV and MV (N=236) | MV Then LJEV (N=235)
Acute bronchitis (Infections and infestations) | 4 | 1 | 5
Acute gastroenteritis (Gastrointestinal disorders) | 8 | 7 | 8
Acute otitis media (Infections and infestations) | 0 | 0 | 1
Acute rhinitis (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 10
Acute Tonsillopharyngitis (Infections and infestations) | 0 | 0 | 1
Atopic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Bacterial conjunctivitis (Infections and infestations) | 1 | 0 | 0
Bronchial asthma (Immune system disorders) | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Enteric fever (Infections and infestations) | 0 | 0 | 1
Impetigo contagious (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Infected wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Insect bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intestinal parasitism (Gastrointestinal disorders) | 0 | 1 | 0
Maculo-papular lesions (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Oral candidiasis (Gastrointestinal disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 1
Post-extraction hematoma (Surgical and medical procedures) | 0 | 1 | 2
Post-vaccination reaction (Surgical and medical procedures) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Roseola infantum (Infections and infestations) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1
Systemic viral infection (Infections and infestations) | 4 | 0 | 2
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 14 | 18 | 42
Viral conjunctivitis (Eye disorders) | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1 | 1
Furuncle (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No